CLINICAL TRIAL: NCT02293018
Title: A Randomized, Single-Blind, Phase 2 Study to Determine the Safety, Tolerability, and Systemic Exposure of 3 Dose Regimens of Topically Applied MTC896 Gel in Subjects With Acne Vulgaris
Brief Title: Pharmacokinetic Study of MTC896 Gel in Subjects With Acne
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mimetica Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MCL14001
Record Dates: First submitted 2014-11-11; First posted 2014-11-18 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.75% (w/w) MTC896 Gel once daily (Experimental): Subjects will apply topically daily 0.75% (w/w) MTC896 Gel
  Interventions: Drug: 0.75% (w/w) MTC896 Gel Once Daily
- 0.75% (w/w) MTC896 Gel twice daily (Experimental): Subjects will apply topically twice daily 0.75% (w/w) MTC896 Gel
  Interventions: Drug: 0.75% (w/w) MTC896 Gel Twice Daily
- 1.5% (w/w) MTC896 Gel once daily (Experimental): Subjects will apply topically daily 1.5% (w/w) MTC896 Gel
  Interventions: Drug: 1.5% (w/w) MTC896 Gel Once Daily

INTERVENTIONS:
Drug: 0.75% (w/w) MTC896 Gel Once Daily
  Arms: 0.75% (w/w) MTC896 Gel once daily
Drug: 0.75% (w/w) MTC896 Gel Twice Daily
  Arms: 0.75% (w/w) MTC896 Gel twice daily
Drug: 1.5% (w/w) MTC896 Gel Once Daily
  Arms: 1.5% (w/w) MTC896 Gel once daily

SUMMARY:
The purpose of this study is to determine the pharmacokinetic properties of topically applied MTC896 Gel following application of 0.75% (w/w) MTC896 Gel once daily and twice daily and 1.5% (w/w) once daily over 4 weeks in the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or nonpregnant female who is at least 18 years of age at the time of screening;
2. Has provided written informed consent (which includes consent for photographs) to be taken at Baseline, EOT, and EOS visits;
3. Has a casual level (CL) of sebum ≥ 150 μg/cm2 on the forehead as measured with the Sebumeter®;
4. Has an SER of ≥ 150 μg/cm2/h on the forehead as measured with the Sebumeter®;
5. Has been diagnosed with inflammatory acne vulgaris of mild to moderate severity defined as:

   * At least 20 inflammatory lesions,
   * At least 20 noninflammatory lesions, and
   * Investigator Global Assessment of 2 or greater;
6. Is willing to comply with the requirements of the protocol;
7. If female and of child-bearing potential, has a negative urine/serum pregnancy test at Screening and Baseline/Day 1 and is willing to use effective contraception during the study. Females are considered to be of childbearing potential unless surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation), diagnosed as infertile, have the same sex partner or a vasectomized male partner, are postmenopausal for at least 1 year, or are abstinent; (Acceptable methods of birth control are defined as: abstinence, oral contraceptives, contraceptive patches/implants; Depo-Provera®, double barrier methods (eg, condom and spermicide) or an IUD. Birth control method must have been stable/unchanged for 12 weeks prior to Baseline and must remain unchanged during study participation);
8. If male, has been vasectomized or agrees to use an accepted method of birth control with female partner during study participation and for 30 days after the last study drug application;
9. Is in good health and free from any disease which, in the opinion of the Investigator, would put the subject at risk if participating in the study;
10. Is free of any systemic or dermatologic disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of adverse events;
11. Is willing to abstain from using any facial treatment products or personal care products (moisturizer, sunscreen, hair spray, etc) on the face during the study;
12. Is willing to avoid sun exposure and to protect the face with a hat/visor;
13. If male, must agree to shave the treatment area and must agree not to alter his routine shaving regimen for the duration of the study;
14. Is willing to refrain from using any treatments, other than the study medication, including antibiotics, for acne present on the face. Topical acne treatments that do not have significant or measurable systemic absorption (eg, benzoyl peroxide, salicylic acid) are allowed for treatment of acne of the back, shoulders, and chest only;

Exclusion Criteria:

1. Pregnant or lactating or plan to become pregnant within 1 month of study completion;
2. Known allergy/sensitivity to any of the drug product components;
3. Any skin condition which may interfere with the evaluation of safety or of acne vulgaris (eg, rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne or folliculitis);
4. Excessive facial hair that would interfere with diagnosis or assessment of acne vulgaris;
5. Excessive sun exposure, in the opinion of the Investigator or, use of tanning booths;
6. Active cystic acne or acne congoblata, acne fulminans, and secondary acne;
7. Two or more active nodular lesions;
8. Screening clinical chemistry or hematology laboratory value that is considered clinically significant, in the opinion of the Investigator;
9. Participation in an investigational drug study within 30 days prior to Screening;
10. Are a poor medical risk because of other systemic diseases or active uncontrolled infections, in the opinion of the Investigator;
11. Any other condition which, in the judgment of the Investigator, would put the subject at unacceptable risk for participation in the study;
12. Treatment with any Cytochrome P450 3A4 (CYP3A4) or Cytochrome P450 3A5 (CYP3A5) inhibitor;
13. Treatment with over-the-counter (OTC) topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid on the face within 2 weeks prior to Baseline;
14. Treatment with systemic corticosteroids (including intranasal and inhaled corticosteroids) within 4 weeks prior to Baseline;
15. Treatment with systemic antibiotics or systemic anti-acne drugs or systemic anti-inflammatory drugs within 4 weeks prior to Baseline;
16. Prescription topical retinoid use on the face within 4 weeks of Baseline (eg, tretinoin, tazarotene, adapalene);
17. Initiation of treatment with hormonal therapy or dose change to hormonal therapy within 12 weeks prior to Baseline. Dose and frequency of use of any hormonal therapy started more than 12 weeks prior to Baseline must remain unchanged throughout the study. Hormonal therapies include, but are not limited to, testosterone, anabolic steroids, and estrogenic and progestational agents such as birth control pills;
18. Use of androgen receptor blockers (such as spironolactone or flutamide) within 3 months prior to Baseline;
19. Oral retinoid use (eg, isotretinoin) within 9 months prior to Baseline or vitamin A supplements greater than 10,000 units/day within 6 months of Baseline;
20. Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 8 weeks or during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic: maximum concentration (Cmax) of MTC896 in the plasma after 28 days of treatment | 4 weeks
  The primary pharmacokinetic outcome measure will be the maximum concentration (Cmax) of MTC896 in the plasma after 28 days of treatment.

SECONDARY OUTCOMES:
Safety and tolerability: Adverse event incidence and severity, local tolerability, laboratory test results, vital signs, 12-lead electrocardiogram | 4 weeks
  Adverse event incidence and severity, local tolerability, laboratory test results (hematology, clinical chemistry, lipid profile, urinalysis), vital signs (systolic and diastolic blood pressure, heart rate, respiratory rate), 12-lead electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - DermResearch, Austin, Texas
  - J&S Studies, College Station, Texas
  - Premier Clinical Research, Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.js-studies.com
- See also: Related Info — http://www.premierclinicalresearch.com